CLINICAL TRIAL: NCT06991023
Title: A Randomised Controlled Trial Exploring the Effects of Prebiotics for Mental Strain and Physiological Markers of Stress in Healthy, Mild-to-Moderately Stressed Adults
Brief Title: Prebiotic Effects on Anxiety, Cortisol, and Emotional Processing in Mild-to-Moderately Stressed Adults
Acronym: PEACE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Clasado Research Services Ltd (Industry)
Responsible Party: Principal Investigator, Daniel Lamport, Associate Professor, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UReading Prebiotics & Stress
Record Dates: First submitted 2025-03-18; First posted 2025-05-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Mild-to-Moderate Stress
Keywords: Randomised Controlled Trial; Stress; Cortisol; Prebiotic
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic (Experimental): The prebiotic supplement (Bimuno®) is a galactooligosaccharide (GOS) supplement derived from lactose which is publicly available and sold in the UK. Subjects will consume a daily dose of 2.75g GOS (3.65g total powder) which will be administered in sachets and consumed with breakfast by mixing into water, tea or coffee, or sprinkling on top of/mixing into food.
  Interventions: Dietary Supplement: Prebiotic (Bimuno®)
- Placebo (Placebo Comparator): The matched placebo contains 3.65g sachets of maltodextrin, and is consumed in the same manner as the prebiotic.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prebiotic (Bimuno®) — The prebiotic supplement (Bimuno®) is a galactooligosaccharide (GOS) supplement derived from lactose which is publicly available and sold in the UK. Subjects will consume a daily dose of 2.75g GOS (3.65g total powder) which will be administered in sachets and consumed with breakfast by mixing into water, tea or coffee, or sprinkling on top of/mixing into food.
  Arms: Prebiotic
Dietary Supplement: Placebo — A matched placebo for the prebiotic intervention, containing 3.65g of maltodextrin. Consumed in the same manner as the prebiotics.
  Arms: Placebo

SUMMARY:
The levels of stress that we experience as a population are continuing to rise due to financial, social and work pressures, particularly in mid-life where additional factors such as family and career often compound these issues. When we experience high levels of stress for prolonged periods, this often has detrimental effects on our mental and physical wellbeing, leading to chronic illness and mental health disorders.

Prebiotics are non-digestible fibres found in food and supplements which promote the growth of beneficial bacteria that produce short-chain fatty acids (SCFAs). Research shows that prebiotics may be used as a lifestyle intervention to support individuals experiencing stress and help reduce physiological and psychological feelings of stress.

As such, this study will build on previous research and explore whether a prebiotic supplement (Bimuno®) has a beneficial effect on stress, mental health outcomes, and sleep in mild-to-moderately stressed adults. To address these questions, participants will take the prebiotic or a placebo for 6 weeks, and visit the University of Reading to complete some questionnaires and cognitive tests at the start and end of the trial. The investigators will also ask participants to collect saliva samples to see if the prebiotics influence cortisol levels, which are linked to stress.

DETAILED DESCRIPTION:
The study employs a parallel groups, randomised, placebo-controlled design in 55 (allowing for 10% attrition) adults aged 25 - 40 experiencing mild-to-moderate stress. Information sheet, consent form, screening and collection of demographic data will be conducted via Redcap at the start of the study. Each participant will then attend 3 in-person sessions at the UoR Psychology department - 1 practice session, and 2 study visits 6 weeks apart. Between the study visits, participants will be required to consume a prebiotic supplement (Bimuno®) once a day at home, and collect saliva samples on 4 occasions.

Screening (all conducted via Redcap) All participants will read through the participant information sheet and sign the consent form before completing a health and lifestyle screening questionnaire to collect demographic data and ensure they meet the eligibility criteria. If eligible, subjects will then be invited to attend an in-person practice visit.

Practice visit The practice visit will be conducted in the Nutrition, Cognition and Health lab in the Psychology department, at any time of day (within working hours) to suit the participant. During this visit, the researcher will double-check participant eligibility and talk the subject through the full trial protocol. Participants will then complete the mood questionnaires and one practice round of the cognitive task (detailed in the study visit section below). This allows participants to see the type of questions they will be asked and ensure they're comfortable answering them, as well as ensure competency on the task before collecting data in the study visits. Finally, participants will be provided with two cycles worth of saliva sample kits and a demonstration on how collect their saliva samples.

Study visit(s) Subjects will consume a standardised breakfast of one slice of white toast and butter with water at home prior to arrival (or, if the participant does not routinely eat breakfast, they may arrive for the visits fasted). Study visits will be conducted in the Nutrition, Cognition and Health lab in the Psychology department, and participants will have the option to arrive anytime between 8am and 11am. This allows participants to complete their study visits before starting their work day if necessary, but also ensures that all sessions are complete before lunch removing the need to provide standardised lunch for participants. Start time of sessions will be kept consistent across visits within participants, as will the choice to have breakfast or not. During the study visits, participants will complete the following mood and sleep questionnaires in a fixed order using Redcap.

Following the questionnaires, participants will complete two emotional cognition tasks in order to explore how the prebiotic supplement might affect emotional processing. All measures will be administered via Inquisit.

At the end of the first study visit, subjects will be provided with their intervention sachets and two more cycles-worth of saliva kits to be used at the end of the study. At the end of the second visit, participants will be given the debrief sheet and emailed a payment form to complete. Both the prebiotic and the matched placebo are supplied by Clasado Research Services Ltd, Reading UK.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25-40
* Meeting at least mildly stressed as per the stress subscale on the Depression, Anxiety and Stress Scale (DASS-42) (score of 15 or more)

Exclusion Criteria:

* Antibiotics within 3 months of enrolment
* Habitual consumption of pre-, pro-, or synbiotics within 3 months of enrolment
* Diagnosis of a mental health disorder within 6 months of enrolment
* Use of antidepressant medication within 6 months of enrolment
* Smoking (defined as having smoked anytime within a month of enrolment
* Following a vegan diet, or dairy or lactose intolerance
* Shift workers with unsocial hours
* Current or historic gastrointestinal disorder, including IBS and IBD
* Current or historic diagnosis of type 1 or 2 diabetes, or any other metabolic disorder
* Current or historic diagnosis of any cardiovascular or related disease/illness
* Current or historic diagnosis of chronic fatigue or cancer
* Current or historic use of weight-loss drugs
* Current of historic diagnosis of any disorder affecting cortisol levels, including Cushing's

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | Baseline
  The PSS is a widely used psychological instrument for measuring the perception of stress. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress. The questions in the PSS ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way using the following 5-point Likert scale: 0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Fairly Often, 4 = Very Often.
Perceived Stress Scale (PSS) | Post-intervention (6 weeks)
  The PSS is a widely used psychological instrument for measuring the perception of stress. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress. The questions in the PSS ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way using the following 5-point Likert scale: 0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Fairly Often, 4 = Very Often.

SECONDARY OUTCOMES:
Positive and Negative Affect Schedule - expanded (PANAS-x) | Baseline
  The PANAS-x is a self-report mood questionnaire measuring overall Positive (PA) and Negative Affect (NA), as well as 11 primary affects including Fear, Sadness, Guilt, Hostility, Shyness, Fatigue, Surprise, Joviality, Self-Assurance, Attentiveness, and Serenity. Participants will be asked to think about how they've been feeling over the past few weeks when using a 5-point Likert scale ranging from 'Very slightly or not at all'; 'A little'; 'Moderately'; 'Quite a bit'; to 'Extremely' to rate each of the 60 adjectives. Scores for the PA and NA subscales range from 0-50. Higher PA scores indicate more positive mood. Higher NA scores indicate more negative mood.
Positive and Negative Affect Schedule - expanded (PANAS-x) | 6 weeks
  The PANAS-x is a self-report mood questionnaire measuring overall Positive (PA) and Negative Affect (NA), as well as 11 primary affects including Fear, Sadness, Guilt, Hostility, Shyness, Fatigue, Surprise, Joviality, Self-Assurance, Attentiveness, and Serenity. Participants will be asked to think about how they've been feeling over the past few weeks when using a 5-point Likert scale ranging from 'Very slightly or not at all'; 'A little'; 'Moderately'; 'Quite a bit'; to 'Extremely' to rate each of the 60 adjectives. Scores for the PA and NA subscales range from 0-50. Higher PA scores indicate more positive mood. Higher NA scores indicate more negative mood.
Patient Health Questionnaire-8 (PHQ-8) | Baseline
  The 8-item version of the Patient Health Questionnaire is a widely used self-report screening questionnaire for depression severity. 8 items are scored using a scale from 8 0 (Not at all) to 3 (Nearly every day), referring to the presence of that symptom during the previous 2 weeks. The PHQ-8 score is the sum of the scores from each of the eight items, and ranges from 0 to 24. Higher scores indicate more severe depression.
Patient Health Questionnaire-8 (PHQ-8) | Post-intervention (6 weeks)
  The 8-item version of the Patient Health Questionnaire is a widely used self-report screening questionnaire for depression severity. 8 items are scored using a scale from 8 0 (Not at all) to 3 (Nearly every day), referring to the presence of that symptom during the previous 2 weeks. The PHQ-8 score is the sum of the scores from each of the eight items, and ranges from 0 to 24. Higher scores indicate more severe depression.
General Anxiety Disorder-7 (GAD-7) | Baseline
  The GAD-7 is a widely used initial screening tool for General Anxiety Disorder, comprising of 7 items which are scored from 0 (not at all) - 3 (nearly every day). Total score for the seven items ranges from 0 to 21, where 0-4: minimal anxiety, 5-9: mild anxiety, 10-14: moderate anxiety, and 15-21: severe anxiety.
General Anxiety Disorder-7 (GAD-7) | Post-intervention (6 weeks)
  The GAD-7 is a widely used initial screening tool for General Anxiety Disorder, comprising of 7 items which are scored from 0 (not at all) - 3 (nearly every day). Total score for the seven items ranges from 0 to 21, where 0-4: minimal anxiety, 5-9: mild anxiety, 10-14: moderate anxiety, and 15-21: severe anxiety.
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  A self-reported measure of sleep quality and disturbances over the past month. Each of the questionnaire's 19 self-reported items belongs to one of seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances.
Pittsburgh Sleep Quality Index (PSQI) | Post-intervention (6 weeks)
  A self-reported measure of sleep quality and disturbances over the past month. Each of the questionnaire's 19 self-reported items belongs to one of seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances.
Salivary Cortisol | 1 day before baseline
  Cortisol (nmol/L), as measured through saliva samples, provides a biomarker of stress, and will be used in the present study to assess whether prebiotic supplementation influences the HPA axis and physiological markers of stress. Saliva samples will be collected in 'sample cycles', with each cycle including 4 time points : 1) before bed, 2) immediately upon waking, 3) 30 minutes after waking, and 4) 45 minutes after waking. Cycles will be collected on two consecutive days at baseline and two consecutive days post-intervention to ensure accurate data.
Salivary Cortisol | Baseline
  Cortisol (nmol/L), as measured through saliva samples, provides a biomarker of stress, and will be used in the present study to assess whether prebiotic supplementation influences the HPA axis and physiological markers of stress. Saliva samples will be collected in 'sample cycles', with each cycle including 4 time points : 1) before bed, 2) immediately upon waking, 3) 30 minutes after waking, and 4) 45 minutes after waking. Cycles will be collected on two consecutive days at baseline and two consecutive days post-intervention to ensure accurate data.
Salivary Cortisol | 1 day before post-intervention measures (6 weeks)
  Cortisol (nmol/L), as measured through saliva samples, provides a biomarker of stress, and will be used in the present study to assess whether prebiotic supplementation influences the HPA axis and physiological markers of stress. Saliva samples will be collected in 'sample cycles', with each cycle including 4 time points : 1) before bed, 2) immediately upon waking, 3) 30 minutes after waking, and 4) 45 minutes after waking. Cycles will be collected on two consecutive days at baseline and two consecutive days post-intervention to ensure accurate data.
Salivary Cortisol | Post-intervention (6 weeks)
  Cortisol (nmol/L), as measured through saliva samples, provides a biomarker of stress, and will be used in the present study to assess whether prebiotic supplementation influences the HPA axis and physiological markers of stress. Saliva samples will be collected in 'sample cycles', with each cycle including 4 time points : 1) before bed, 2) immediately upon waking, 3) 30 minutes after waking, and 4) 45 minutes after waking. Cycles will be collected on two consecutive days at baseline and two consecutive days post-intervention to ensure accurate data.
Epic-Norfolk Food Frequency Questionnaire | Baseline
  The FFQ is a validated tool for gauging the average habitual dietary intake of micro and macronutrients of an individual in the UK. Data will be processed using the FETA software.
FibreScreen | Baseline
  A short fibre screening questionnaire, the 18-item FiberScreen was developed and validated to reduce the burden of dietary screening of fibre intake for both participant and researcher. The FiberScreen includes questions about fruits, dried fruits, vegetables, bread, whole grain, pasta/rice/potato, legumes and nuts and seeds intake of the last 2 weeks.
FibreScreen | Post-intervention (6 weeks)
  A short fibre screening questionnaire, the 18-item FiberScreen was developed and validated to reduce the burden of dietary screening of fibre intake for both participant and researcher. The FiberScreen includes questions about fruits, dried fruits, vegetables, bread, whole grain, pasta/rice/potato, legumes and nuts and seeds intake of the last 2 weeks.
Emotion dot probe task | Baseline
  A cognitive task which is used to measure attentional biases towards emotional stimuli. Participants respond to a probe (letter) appearing in the location of either a neutral or emotional word. Faster responses when the probe appears in the location of the emotional stimulus indicates a bias towards the emotional stimulus. Outcome measures include: accuracy when probe is presented in position of negative stimuli (negative trial, congruent); accuracy when probe is presented in position of neutral stimuli (negative trial, incongruent); accuracy when probe is presented in position of positive stimuli (positive trial, congruent); accuracy when probe is presented in position of neutral stimuli (positive trial, incongruent); RT for negative congruent & incongruent; RT for positive congruent & incongruent; negative attentional bias; positive attentional bias.
Emotion dot probe task | Post-intervention (6 weeks)
  A cognitive task which is used to measure attentional biases towards emotional stimuli. Participants respond to a probe (letter) appearing in the location of either a neutral or emotional word. Faster responses when the probe appears in the location of the emotional stimulus indicates a bias towards the emotional stimulus. Outcome measures include: accuracy when probe is presented in position of negative stimuli (negative trial, congruent); accuracy when probe is presented in position of neutral stimuli (negative trial, incongruent); accuracy when probe is presented in position of positive stimuli (positive trial, congruent); accuracy when probe is presented in position of neutral stimuli (positive trial, incongruent); RT for negative congruent & incongruent; RT for positive congruent & incongruent; negative attentional bias; positive attentional bias.
Emotion Go/No-Go task | Baseline
  A go/no-go task where participants press the spacebar to respond to 'go' trials and withhold pressing the spacebar on 'no-go' trials, measuring inhibitory control and attention. This task contains 8 conditions which are presented in a random order: Fear Go, Neutral No-Go; Neutral Go, Fear No-Go; Happy Go, Neutral No-Go; Neutral Go, Happy No-Go; Sad Go, Neutral No-Go; Neutral Go, Sad No-Go; Angry Go, Neutral No-Go; Neutral Go, Angry No-Go. Outcome measures include hit rate (correctly responding to go trails), miss rate (1 - hit rate), overall commission error (pressing space on no-go), rejection rate (1-commission error), hit reaction time. Each of these outcome measures is also calculated per emotional condition.
Emotion Go/No-Go task | Post-intervention (6 weeks)
  A go/no-go task where participants press the spacebar to respond to 'go' trials and withhold pressing the spacebar on 'no-go' trials, measuring inhibitory control and attention. This task contains 8 conditions which are presented in a random order: Fear Go, Neutral No-Go; Neutral Go, Fear No-Go; Happy Go, Neutral No-Go; Neutral Go, Happy No-Go; Sad Go, Neutral No-Go; Neutral Go, Sad No-Go; Angry Go, Neutral No-Go; Neutral Go, Angry No-Go. Outcome measures include hit rate (correctly responding to go trails), miss rate (1 - hit rate), overall commission error (pressing space on no-go), rejection rate (1-commission error), hit reaction time. Each of these outcome measures is also calculated per emotional condition.
Gastrointestinal Symptoms Rating Scale (GSRS) | Post-intervention (6 weeks)
  A 15-item questionnaire to ascertain whether participants experienced any gastrointestinal side effects of consuming either the prebiotic or placebo. Participants will also be asked whether the level of experience they report for each symptom is better than, worse than, or the same as prior to taking part in the trial

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lamport, PhD, Principal Investigator — University of Reading; Piril Hepsomali, Study Director — University of Reading; Claire Williams, Study Director — University of Reading
Locations (1):
- Nutrition, Cognition & Health Lab, School of Psychology and Clinical Language Sciences, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All questionnaire, cognitive, and saliva data will be preserved and may be made available in anonymised form on a public repository such as the University of Reading Research Data Archive at the end of the project, in accordance with Open Science Principles.